CLINICAL TRIAL: NCT06233006
Title: Investigation of the Effects of Upper Extremity Functions and Health-Related Quality of Life in Female Patients With Non-Specific Neck Pain
Brief Title: Investigation of the Effects of Upper Extremity Functions in Female Patients With Non-Specific Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: Tarsus University (Other)
Responsible Party: Principal Investigator, Abdulkadir GOZ, MsC, Dokuz Eylul University
Other Study IDs: DokuzEU01
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non Spesific Neck Pain: Patients with Non Spesific Neck Pain
  Interventions: Other: Assessment
- Healthy Control: Individuals with similar age
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — upper extremity functions (hand skills, hand and finger grip strength, reaction time, position sense, upper extremity strength and endurance) and health-related quality of life

SUMMARY:
Non-specific neck pain is defined as pain in the posterior and lateral part of the neck between the superior nuchael line and the spinous process of the 1st thoracic vertebra, without neurological findings and obvious structural pathology. It is more common in women than in men. Neck pain is thought to affect upper extremity functions. Although the exact cause is unknown, it has been reported that mechanical loading, minor peripheral nerve damage and deconditioning negatively affect upper extremity functions in individuals with neck pain and reduce the quality of life. Although it is stated in the literature that patients with neck pain often experience upper extremity problems, there are a limited number of studies evaluating the relationship between the neck and upper extremity.

This study was planned to determine upper extremity functions and their impact on health-related quality of life in female patients with NSHP. Female patients with NSHP over the age of 18 who apply to Tarsus State Hospital Physical Therapy and Rehabilitation Clinic, meet the inclusion criteria, and agree to participate in the study will be included in the study. With our research, patients' upper extremity functions (hand skills, hand and finger grip strength, reaction time, position sense, upper extremity strength and endurance) and health-related quality of life will be evaluated and interpreted.

DETAILED DESCRIPTION:
Non-specific neck pain is defined as pain in the posterior and lateral part of the neck between the superior nuchael line and the spinous process of the 1st thoracic vertebra, without neurological findings and obvious structural pathology. It is more common in women than in men. Neck pain is thought to affect upper extremity functions. Although the exact cause is unknown, it has been reported that mechanical loading, minor peripheral nerve damage and deconditioning negatively affect upper extremity functions in individuals with neck pain and reduce the quality of life. Although it is stated in the literature that patients with neck pain often experience upper extremity problems, there are a limited number of studies evaluating the relationship between the neck and upper extremity.

This study was planned to determine upper extremity functions and their impact on health-related quality of life in female patients with NSHP. Female patients with NSHP over the age of 18 who apply to Tarsus State Hospital Physical Therapy and Rehabilitation Clinic, meet the inclusion criteria, and agree to participate in the study will be included in the study. With our research, patients' upper extremity functions (hand skills, hand and finger grip strength, reaction time, position sense, upper extremity strength and endurance) and health-related quality of life will be evaluated and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain lasting more than 30 days and being diagnosed with non-specific neck pain
* Having a score of 14/50 or above on the Neck Disability Index
* Expressing neck pain as at least 3/10 points or above on the visual analog scale
* Being 18 years or older
* Female patients

Exclusion Criteria:

* Previously diagnosed orthopedic diseases related to the spine
* Undergoing surgical upper extremity surgery that may affect upper extremity functions
* Being pregnant and having just given birth
* Serious pathologies (such as cancer, spondylolisthesis, rheumatoid arthritis, kyphoscoliosis, scoliosis, etc., thoracic deformity or ankylosing spondylitis)
* Symptoms of cervical spinal stenosis (such as incoordination of hands, arms and legs, bowel and bladder incontinence)
* Radix compression (such as sensory changes, muscle weakness, or decreased reflexes)
* History of whiplash or cervical surgery
* Kyphoscoliosis, scoliosis etc. thorax deformity
* Having a body mass index over 30

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with Non Spesific Neck Pain
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
hand skills | 4 minutes
  Assessed with Nine Hole Peg Test
hand grip strength | 1 minute
  Assessed with Baseline Hand Dynamometer
pinch grip strength | 1 minute
  Assessed with Baseline Pinchmeter
reaction time | 1 minute
  Assessed with Nelson Hand Reaction Test
position sense | 5 minutes
  Assessed with Baseline Digital Inclinometer
Upper extremity strength and endurance | 1 minutes
  Assessed with Single Arm Military Press Test
upper extremity disability | 5 minutes
  Assessed with DASH questionnarie

SECONDARY OUTCOMES:
Health Related Quality of Life | 5 minutes
  Assessed with SF36 quastionnarie
Neck disability | 5 minutes
  Assessed with Neck Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi OZALEVLİ, PhD, Study Director — Dokuz Eylul University
Locations (1):
- Tarsus State Hospital, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No